CLINICAL TRIAL: NCT02637453
Title: Addition of Six Short Ablation Lines on Pulmonary Vein Isolation Circumferences Reduces Recurrence Rate of Paroxysmal Atrial Fibrillation
Brief Title: Addition of Six Short Lines on Pulmonary Vein Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xuzhou Central Hospital (Other); Shanghai East Hospital (Other); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Yi-Gang Li, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiXinhua-Af
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI (Active Comparator): Pulmonary vein isolation (PVI)
  Interventions: Procedure: PVI
- PVI+6L (Experimental): PVI plus 6 additional lines at 1, 3 and 6 o'clock (from internal view) of left PV and 6, 9 and 11 o'clock of right PV
  Interventions: Procedure: CPVI+6L

INTERVENTIONS:
Procedure: PVI — Pulmonary vein isolation
  Arms: PVI
Procedure: CPVI+6L — After PVI, 6 ablation lines were added with an extension from pulmonary vein ostium at 1, 3 and 6 o'clock (from internal view) of left PV and 6, 9 and 11 o'clock of right PV
  Arms: PVI+6L

SUMMARY:
We randomly assigned 390 patients with symptomatic, paroxysmal AF to undergo catheter ablation with PVI (PVI group) alone or combined with 6 additional ablation lines extended outside the PVI circumferences at 1, 3 and 6 o'clock of left PV and 6, 9 and 11 o'clock of right PV (PVI+6L group). Patients received monthly 12-lead electrocardiogram, 24-hour Holter at 3, 6 and 9 months and 14-days continuous monitoring at 12 months to detect atrial tachyarrhythmia. The follow-up period was 12 months. The primary end point was freedom from AF recurrence between 91 and 365 days after catheter ablation. The secondary end points included the AF burden, procedural parameters, and complications.

DETAILED DESCRIPTION:
We randomly assigned 390 patients with symptomatic, paroxysmal AF to undergo catheter ablation with PVI (PVI group) alone or combined with 6 additional ablation lines extended outside the PVI circumferences at 1, 3 and 6 o'clock of left PV and 6, 9 and 11 o'clock of right PV (PVI+6L group). Patients received monthly 12-lead electrocardiogram, 24-hour Holter at 3, 6 and 9 months and 14-days continuous monitoring at 12 months to detect atrial tachyarrhythmia. The follow-up period was 12 months. The primary end point was freedom from AF recurrence between 91 and 365 days after catheter ablation. The secondary end points included the AF burden, procedural parameters, and complications.

ELIGIBILITY:
Inclusion criteria

1. Patients between the ages of 18 and 80 years undergoing their first ablation of atrial fibrillation.
2. Diagnosed with symptomatic paroxysmal atrial fibrillation, defined as an documented episode of atrial fibrillation that lasts more than 30 seconds and terminates in less than 7 days.
3. Resistant or intolerant to at least one class I, II, or III antiarrhythmic drugs.
4. Patients deemed candidates for radiofrequency ablation of atrial fibrillation.
5. Able and willing to comply with pre-, post-, and follow-up requirements.

Exclusion criteria

1. Left atrial thrombus by pre-procedural imaging.
2. Uncontrolled heart failure: New York Heart Association Class III or IV, or left ventricular ejection fraction< 40%
3. Myocardial infarction, unstable angina, coronary stenting within the previous 90 days.
4. Stroke or any thrombo-embolic events within the previous 90 days.
5. Expecting cardiac transplantation or other cardiac surgery within 180 days.
6. History of catheter ablation of atrial fibrillation, atrial flutter or atrial tachycardia.
7. History of blood clotting or bleeding abnormalities.
8. Contraindication to anticoagulation.
9. History of cardiac surgery.
10. Uncontrolled maligment tumor.
11. Patients in dialysis or creatinine > 221 μmol/L.
12. Patients with alanine aminotransferase > 150 U/L or aspartate aminotransferase > 76 U/L
13. Acute illness or active infection at time of index procedure or leukocytosis for which antibiotics have been or will be prescribed.
14. Life expectancy less than 1 year.
15. Women who are pregnant or who plan to become pregnant during the study.
16. Other significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Freedom from AF recurrence between 91 and 365 days | 91 to 365 days
  AF recurrence was defined by AF (including atrial flutter or atrial tachycardia) of 30 seconds or more captured by ECG monitoring or any clinical presentation with AF outside the 90-day blanking period (between 91 and 365 days). Cardioversion, or use of class I or III antiarrhythmic drugs outside blanking period was also considered as AF recurrence.

SECONDARY OUTCOMES:
AF burden | 12 months
  Percentage of time in AF, atrial flutter or atrial tachycardia on 14-days continuous monitoring at 12 months.
Procedural time | Within procedure
  Total procedural time from femoral vein puncture to decannulation (skin-to-skin time)
Fluoroscopy time | Within procedure
  Time of patients' exposure to the real-time X-ray imaging during the procedure.
Ablation time | Within procedure
  Radiofrequency delivery time during the procedure.
Early onset complications | Within 30 days
  Complications within 30 days post-ablation, including death, myocardial infarction, diaphragmatic paralysis, stroke or transient ischemic attack, systemic embolism, pericardial effusion or tamponade requiring drainage, heart block, pericarditis, and vascular access complications requiring intervention.
Late onset complications | within 12 months
  Complications detected any time during the follow-up, including severe pulmonary vein stenosis (>70%), and atrioesophageal fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, MD., Principal Investigator — Department of Cardiology, Xinhua Hospital, Shanghai Jiaotong University School of Medicne
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicne, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Steinberg BA, Beckley PD, Deering TF, Clark CL, Amin AN, Bauer KA, Cryer B, Mansour M, Scheiman JM, Zenati MA, Newby LK, Peacock WF, Bhatt DL; Society of Cardiovascular Patient Care. Evaluation and management of the atrial fibrillation patient: a report from the Society of Cardiovascular Patient Care. Crit Pathw Cardiol. 2013 Sep;12(3):107-15. doi: 10.1097/HPC.0b013e31829834ed. PMID 23892939
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Zhang S. Atrial fibrillation in mainland China: epidemiology and current management. Heart. 2009 Jul;95(13):1052-5. doi: 10.1136/hrt.2008.146589. Epub 2009 Mar 23. PMID 19318342
- [Background] Weerasooriya R, Khairy P, Litalien J, Macle L, Hocini M, Sacher F, Lellouche N, Knecht S, Wright M, Nault I, Miyazaki S, Scavee C, Clementy J, Haissaguerre M, Jais P. Catheter ablation for atrial fibrillation: are results maintained at 5 years of follow-up? J Am Coll Cardiol. 2011 Jan 11;57(2):160-6. doi: 10.1016/j.jacc.2010.05.061. PMID 21211687
- [Background] Cheema A, Vasamreddy CR, Dalal D, Marine JE, Dong J, Henrikson CA, Spragg D, Cheng A, Nazarian S, Sinha S, Halperin H, Berger R, Calkins H. Long-term single procedure efficacy of catheter ablation of atrial fibrillation. J Interv Card Electrophysiol. 2006 Apr;15(3):145-55. doi: 10.1007/s10840-006-9005-9. Epub 2006 Aug 5. PMID 17019636
- [Background] Ouyang F, Tilz R, Chun J, Schmidt B, Wissner E, Zerm T, Neven K, Kokturk B, Konstantinidou M, Metzner A, Fuernkranz A, Kuck KH. Long-term results of catheter ablation in paroxysmal atrial fibrillation: lessons from a 5-year follow-up. Circulation. 2010 Dec 7;122(23):2368-77. doi: 10.1161/CIRCULATIONAHA.110.946806. Epub 2010 Nov 22. PMID 21098450
- [Background] Calo L, Rebecchi M, Sciarra L, De Luca L, Fagagnini A, Zuccaro LM, Pitrone P, Dottori S, Porfirio M, de Ruvo E, Lioy E. Catheter ablation of right atrial ganglionated plexi in patients with vagal paroxysmal atrial fibrillation. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):22-31. doi: 10.1161/CIRCEP.111.964262. Epub 2011 Dec 6. PMID 22147839
- [Background] Katritsis DG, Pokushalov E, Romanov A, Giazitzoglou E, Siontis GC, Po SS, Camm AJ, Ioannidis JP. Autonomic denervation added to pulmonary vein isolation for paroxysmal atrial fibrillation: a randomized clinical trial. J Am Coll Cardiol. 2013 Dec 17;62(24):2318-25. doi: 10.1016/j.jacc.2013.06.053. Epub 2013 Aug 21. PMID 23973694
- [Background] Noheria A, Kumar A, Wylie JV Jr, Josephson ME. Catheter ablation vs antiarrhythmic drug therapy for atrial fibrillation: a systematic review. Arch Intern Med. 2008 Mar 24;168(6):581-6. doi: 10.1001/archinte.168.6.581. PMID 18362249
- [Background] Stabile G, Bertaglia E, Senatore G, De Simone A, Zoppo F, Donnici G, Turco P, Pascotto P, Fazzari M, Vitale DF. Catheter ablation treatment in patients with drug-refractory atrial fibrillation: a prospective, multi-centre, randomized, controlled study (Catheter Ablation For The Cure Of Atrial Fibrillation Study). Eur Heart J. 2006 Jan;27(2):216-21. doi: 10.1093/eurheartj/ehi583. Epub 2005 Oct 7. PMID 16214831
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733